CLINICAL TRIAL: NCT06030193
Title: A Randomized, Active-controlled, Multi-site, Double-masked, Pilot Study to Evaluate the Safety and Tolerability of QLS-111 Versus Timolol Maleate Preservative Free 0.5% Ophthalmic Solution in Subjects With Normal Tension Glaucoma (NTG)
Brief Title: Study of an Investigational Product, QLS-111, Provided as an Eyedrop, for Treatment of Normal Tension Glaucoma (NTG)
Acronym: Nightingale
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qlaris Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QC-111-202; Nightingale (Other: Qlaris Bio, Inc.)
Record Dates: First submitted 2023-08-18; First posted 2023-09-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Normal Tension Glaucoma (NTG); Low-Tension Glaucoma, Bilateral; Low-Tension Glaucoma, Unspecified Eye; Glaucoma
Keywords: NTG; Qlaris; intraocular pressure (IOP); Glaucoma; Nightingale; low-tension glaucoma
MeSH Terms: conditions — Low Tension Glaucoma; Glaucoma | interventions — Ophthalmic Solutions; Timolol

STUDY DESIGN:
Intervention Model Description: Multi site double masked, active-controlled, randomized, prospective parallel, pilot study of 7 days' QPM dosing, followed by 7 days' BID dosing (7 days of dosing per regimen [14-day treatment period]) of an investigational product (IP), QLS-111 or Timolol. Both eyes (OU) will be dosed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study subjects, Investigators and their staff, and Sponsor personnel involved with the conduct and monitoring of the study will be masked to the IP identity until after the final database is locked. IP will be provided in identical appearing packaging. Unmasked statistician preparing the masked randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QLS-111 ophthalmic solution (Experimental): Qlaris' investigational product, QLS-111 ophthalmic solution, 0.15%, provided in single use vials, masked, and PF.
  Interventions: Drug: QLS-111 ophthalmic solution (0.015%)
- Timolol maleate PF 0.5% Ophthalmic Solution (Active Comparator): Timolol BID: Timolol Maleate PF 0.5% Ophthalmic Solution (Timolol) provided in single use vials, masked.
  Interventions: Drug: Timolol Maleate PF 0.5% Ophthalmic Solution (Timolol)

INTERVENTIONS:
Drug: QLS-111 ophthalmic solution (0.015%) — QLS-111 ophthalmic solution 0.015% applied QPM OU for 7 days followed by BID dosing OU for 7 days, to constitute a 14-day study treatment period. All IP for this study will be supplied masked in PF single use vials.
  Other Names: QLS-111
  Arms: QLS-111 ophthalmic solution
Drug: Timolol Maleate PF 0.5% Ophthalmic Solution (Timolol) — Timolol BID: Timolol Maleate PF 0.5% Ophthalmic Solution (Timolol) with BID dosing OU will be administered up to 14 days. All IP for this study will be supplied masked in PF single use vials.
  Other Names: Timolol
  Arms: Timolol maleate PF 0.5% Ophthalmic Solution

SUMMARY:
Qlaris' Phase 2 clinical trial investigating the safety, tolerability, and ocular hypotensive efficacy of QLS-111 in normal tension glaucoma patients.

DETAILED DESCRIPTION:
A randomized, active-controlled, multi-site, double-masked, pilot study to evaluate the safety and tolerability of QLS-111 0.015% versus Timolol maleate ophthalmic preservative free (PF) 0.5% ophthalmic solution in subjects with NTG. Primary objective is to evaluate the ocular and systemic safety and tolerability of QLS-111 0.015% compared to active control (Timolol).

Secondary objective is to evaluate the ocular hypotensive efficacy of QLS-111 0.015% with once daily evening (QPM) and twice daily (BID) dosing versus Timolol with QPM dosing.

ELIGIBILITY:
Inclusion Criteria:

* 30 years or older
* Able to provide written acknowledgement of giving informed consent
* Best corrected visual acuity (BCVA) 20/200 or better
* NTG in both eyes with untreated IOP <21 mmHg at Visit 2 and morning assessment of Visit 3; IOP at morning assessment on Visits 2 and 3 doesn't differ more than 2 mmHg; has open iridocorneal angles, historic IOP <22 mmHg in either eye

Exclusion Criteria:

* History of angle closure glaucoma, narrow or occludable angle on gonioscope
* All secondary glaucomas
* Severe glaucomatous damage that would preclude safe washout of prescribed ocular hypotensive medications
* Previous glaucoma surgery, certain procedures (trabeculotomy, shunt/tubes, cyclodestructive procedure) (selective laser trabeculoplasty (SLT) allowed if done no earlier than 1 year from study, some minimally invasive glaucoma surgeries are allowed if done no earlier than 1.5 years from study)
* Ocular trauma, ocular infections, ocular inflammation, herpes simplex keratitis of eye
* Use of other ophthalmic concomitant medications during the study
* Refractive surgery
* Uncontrolled hypertension or hypotension
* Significant systemic or psychiatric disease
* Participation in other investigational trial 30 days prior to screening or previous enrollment and treatment with Qlaris investigational product
* Pregnant or lactating

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular symptoms and ocular treatment-emergent adverse events (TEAEs) | 14 days
  Ocular safety and tolerability: (AEs)
Clinically significant change in visual acuity | 14 days
  Ocular safety and tolerability: visual acuity
Clinically significant change in findings on slit lamp exam | 14 days
  Ocular safety and tolerability: dilated biomicroscopy of eye to observe clinically significant changes from baseline
Clinically significant change in findings on fundus exam | 14 days
  Ocular safety and tolerability: dilated ophthalmoscopy to observe clinically significant changes from baseline in posterior segment of eye
Incidence of systemic TEAEs | 14 days
  Systemic safety and tolerability: AEs
Clinically significant changes in blood pressure (BP) | 14 days
  Systemic safety and tolerability: vital sign, measuring systolic and diastolic blood pressure
Clinically significant changes in heart rate (HR) | 14 days
  Systemic safety and tolerability: vital signs

SECONDARY OUTCOMES:
Change from baseline (CFB) of diurnal intraocular pressure (IOP) in the study eye | 14 days
  Ocular hypotensive efficacy: diurnal IOP CFB
CFB in IOP at various timepoints in the study eye | 14 days
  Ocular hypotensive efficacy: IOP CFB for multiple timepoints throughout the day

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brandano, Study Director — Qlaris Bio, Inc.
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website, pipeline — https://qlaris.bio